CLINICAL TRIAL: NCT04652076
Title: A Randomized, Multicenter, Open Label, Phase I/II Study to Evaluate the Safety, Clinical and Biological Activity of a Humanized Monoclonal Antibody Targeting Netrin-1 (NP137) in Combination with Carboplatin Plus Paclitaxel And/or Pembrolizumab in Patients with Locally Advanced/metastatic Endometrial Carcinoma or Cervix Carcinoma Progressing/relapsing After At Least One Prior Systemic Chemotherapy.
Brief Title: GYNecological Cancers Treated with NETrin MAbs in Combination with Chemotherapy and /or Pembrolizumab
Acronym: GYNET
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NETRIS Pharma (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP137CT02; 2020-000172-38 (EudraCT Number); /ET20-049 (Other: Centre Léon Berard protocol number); ANR-18-RHUS-0009 (Other Grant/Funding Number: Agence Nationale de Recherche); KEYNOTE-A92 (Other: Merck Sharp & Dohme Corp. protocol number)
Record Dates: First submitted 2020-11-05; First posted 2020-12-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Endometrial Carcinoma; Cervix Carcinoma
Keywords: anti-Netrin 1; anti-PD-1; Immunotherapy; Check Point Inhibitors; Dependence Receptors
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — netrin-1 inhibitor NP137; pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A: Standard Chemotherapy alone (Paclitaxel + Carboplatin) (Other): Standard Chemotherapy will be adminitred in 2 independant cohorts: Endometrial carcinoma or Cervix Carcinoma
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Arm B: Experimental double combination [Standard Chemotherapy +NP137] (Other): Experimental double combination [Standard Chemotherapy +NP137] will be administred in 2 independant cohorts: Endometrial carcinoma or Cervix Carcinoma
  Interventions: Drug: NP137; Drug: Paclitaxel; Drug: Carboplatin
- Arm C: Experimental double combination [Pembrolizumab +NP137] (Other): Experimental double combination [Pembrolizumab +NP137] will be administred in 2 independant cohorts: Endometrial carcinoma or Cervix Carcinoma
  Interventions: Drug: NP137; Drug: Pembrolizumab
- Arm D: Experimental triple therapeutical combination [Pembrolizumab+ Standard Chemotherapy + NP137] (Other): Experimental triple combination [Pembrolizumab+ Standard Chemotherapy + NP137] will be administred in 2 independant cohorts: Endometrial carcinoma or Cervix Carcinoma
  Interventions: Drug: NP137; Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: NP137 — Recombinant humanized IgG1 monoclonal antibody against Netrin 1. NP137 will be administred IV, Q3W until disease progression, unacceptable toxicity, death, patient or physician decision to withdraw, pregnancy or SMPC guidance, whichever occurs first.
  Arms: Arm B: Experimental double combination [Standard Chemotherapy +NP137]; Arm C: Experimental double combination [Pembrolizumab +NP137]; Arm D: Experimental triple therapeutical combination [Pembrolizumab+ Standard Chemotherapy + NP137]
Drug: Pembrolizumab — Humanised monoclonal anti-programmed cell death-1 (PD-1) antibody will be administred in IV Q3W. A maximum 35 cycles of treatments (approximately 2 years) with pembrolizumab can be administered to patients.
  Other Names: KEYTRUDA
  Arms: Arm C: Experimental double combination [Pembrolizumab +NP137]; Arm D: Experimental triple therapeutical combination [Pembrolizumab+ Standard Chemotherapy + NP137]
Drug: Paclitaxel — Standard Chemotherapy agent will be administred IV, Q3W, up to 6 cycles of treatment.
  Arms: Arm A: Standard Chemotherapy alone (Paclitaxel + Carboplatin); Arm B: Experimental double combination [Standard Chemotherapy +NP137]; Arm D: Experimental triple therapeutical combination [Pembrolizumab+ Standard Chemotherapy + NP137]
Drug: Carboplatin — Standard Chemotherapy agent will be administred IV, Q3W, up to 6 cycles of treatment.
  Arms: Arm A: Standard Chemotherapy alone (Paclitaxel + Carboplatin); Arm B: Experimental double combination [Standard Chemotherapy +NP137]; Arm D: Experimental triple therapeutical combination [Pembrolizumab+ Standard Chemotherapy + NP137]

SUMMARY:
The aim of this study is to investigate the safety and the clinical activities of NP137 when combined with pembrolizumab and/or chemotherapies in patients with advanced/metastatic gynecological cancers (2 types: endometrial carcinoma and cervix carcinoma).

DETAILED DESCRIPTION:
The prognosis of patients with locally advanced/metastatic uterine (endometrial or cervical) cancer progressing/relapsing after at least one prior systemic treatment remains poor. The development of new innovative anti-tumor drug candidates as single agent or in combination with chemotherapy or check point inhibitors is needed.

NP137 is a first-in-class humanized monoclonal antibody targeting specifically and selectively Netrin-1. By blocking Netrin-1, NP137 is capable of restoring apoptosis in tumor cells in vitro and in vivo, leading to therapeutic activity in various animal cancer models.

Dependence receptors inhibitor such as NP137 might be a novel choice to improve the clinical outcomes of these patients.

The herein proposed study will be a multicenter, open-label, randomized, Phase I/II trial with:

A safety run in part to assess the safety of the therapeutic combinations for the first 6 patients enrolled in each of the therapeutic combinations independently of the tumor type. According to safety rules, these therapeutic combinations will be investigated or not in the Phase II part.

A Phase II part will be then conducted using an adaptive Bayesian approach allowing to quickly stop treatment cohorts without evidence of efficacy and/or select promising treatment cohorts. The Phase II part will be initiated with a preliminary step to assess the clinical activity of the proposed therapeutic combinations in 2 tumor types before proceeding to the activation of extension phase II part of the study. For each cohorts, clinical activity will be assessed through by sequential statistical analysis at specific timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Be women ≥ 18 years at time of inform consent signature.
* Patient with histologically confirmed locally advanced / metastatic endometrial carcinoma (Endometrial sarcoma are excluded) or patient with histologically confirmed locally advanced / metastatic cervix adeno- or epidermoid- carcinoma.
* Previously treated by at least one line of platinum based chemotherapy, but no more than 3 lines of chemotherapies whatever the nature. If the previous based platinum chemotherapy was given as neoadjuvant or adjuvant chemotherapy for a local disease (stage I or II), inclusion must be performed no more than one year after the end of this chemotherapy, except if an advanced or metastatic relapse has been documented and treated by a systemic anti-cancer agent during this time interval.

In all cases, a minimal wash-out period of 6 months after completion of last chemotherapy with [platinum + paclitaxel] is required prior to entering the study.

Platinum chemotherapy concomitant to RT can not be considered as a line of previous platinum based chemotherapy.

* For endometrium carcinoma: mutational profile (MSI/MSS status) available before randomization (see St Paul de Vence 2019- ARCAGY - GINECO Group recommendation).
* Documented disease progression as per RECIST V1.1 after prior systemic chemotherapy regimen and presence of at least one lesion evaluable for response according to RECIST 1.1.
* Have provided a representative archival tumor sample in formalin-fixed paraffin embedded (FFPE) block (primary tumor or metastasis) or newly obtained core or excisional biopsy of a tumor lesion together with an associated pathology report.

Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut (details pertaining to tumor tissue submission can be found in the laboratory manual).

- Optional for patients having consented to tumor biopsies: presence of at least one tumor lesion visible by medical imaging and accessible to repeatable percutaneous sampling that permits core needle biopsy without unacceptable risk of a significant procedural complications, and suitable for retrieval of 4 cores using a 16-gauge diameter needle or larger.

Note: lesions to be biopsied should not be selected as RECIST target lesions. Bone lesions are not adequate lesions for biopsies and lymph nodes lesions should not be considered as prime targets.

* Life expectancy ≥ 3 months.
* Eastern Cooperative Oncology GrougGroup performance status (ECOG PS) of 0 to 1.
* Demonstrate adequate cardiovascular function:

  * QTcF < 470ms
  * Resting BP systolic <160mmHg and diastolic < 100mmHg
  * LVEF > 50% as determined by transthoracic echocardiogram.
* Demonstrate adequate organ function as defined in protocol, all screening laboratory tests should be performed within 7 days prior C1D1:
* Women of child-bearing potential must have a negative urine pregnancy test at screening (within 72 hours prior C1D1) and must agree to use 2 effective forms of contraception from the time of the treatment period and of the negative pregnancy test up 6 months after the end of their treatment.
* Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures.
* Patient should be able and willing to comply with study visits and procedures as per protocol.

Exclusion Criteria:

* Patients with progression during previous chemotherapy with [platinum +paclitaxel]
* Persistence of CTCAE ≥ Grade 2 toxicity due to prior anti-cancer therapy (except alopecia (any grades).
* History of severe (≥Grade 3) allergic anaphylactic reactions to one of the components of NP137, pembrolizumab, paclitaxel, carboplatin and/or any of their excipients.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years.

Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

* Prior/concomitant Therapy:

  * Have received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade ≥ 3 irAE
  * Have received prior systemic anti-cancer therapy :
* Chemotherapy or targeted therapies (approved or investigational) within 2 weeks or 5* t1/2 whichever is longer prior C1D1.
* Hormonal therapy within 1 week prior to C1D1
* Biological therapy within 4 weeks prior to C1D1

  * Are currently participating in or have participated in a study of an investigational agent or have used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent. Have received prior radiotherapy within 4 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
  * Have had major surgery within 4 weeks of start of study treatment. Participants must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment, C1D1.
  * Have received a live or live-attenuated vaccine within 30 days prior to the first dose of study drug. Note: killed vaccinesare allowed.
  * Have received immunosuppressive medication within 2 weeks with the exceptions of intranasal, topical and inhaled corticosteroids or systemic corticosteroids at doses which are not to exceed 10 mg/day of prednisone, or equivalent doses of another corticosteroid.
* Have a history of autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed. History of autoimmune disease which include but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on stable thyroid replacement hormone therapy,
  * Patients with controlled Type 1 diabetes mellitus,
  * patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are eligible provided that they meet the following conditions:

    * Rash must cover less than 10% of body surface area (BSA).
    * Disease is well controlled at baseline and only requiring low potency topical steroids.
    * No acute exacerbations of underlying condition within the previous 12 months requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoid, biologic agents, oral calcineurin inhibitors, high potency or oral steroids.
* Patients with HIV, active B or C hepatitis infection. Notes: Active hepatitis B i.e. chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening before C1D1. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to C1D1. Patients with a positive HBcAb test must have a negative HBV DNA test at screening. Active hepatitis C i.e. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA at screening.
* Patients with active tuberculosis.
* Prior allogeneic bone marrow transplantation or solid organ transplant for another malignancy in the past.
* History of idiopathic pulmonary fibrosis, non-infectious pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease , drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.
* Have an active infection requiring systemic therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
DLT occurrence | Safety run in Period: At the end of Cycle 2 (each cycle is 21 days) for the first 6 to 12 patients per arm
  Any pre-definied toxicities graded by using NCI CTCAE Version 5.0 and assessed by the investigator to be possibly, probably, or definitely related to study treatments administration during the safety run in period
Overall response Rate (ORR) | At 3 months of treatement and then every 12 weeks, up to 2 years
  Rate of patients with CR or PR as per RECIST 1.1

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Every 12 weeks, up to 2 years
  The proportion of evaluable patients with an objective response according to RECIST 1.1.
Duration of Response | Every 12 weeks, up to 2 years
  Time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the first date that disease progression or death is documented,
Progression-free Survival | Every 12 weeks, up to 2 years
  Time from first study drug intake until disease progression or death, whichever occurs first
Overall Survival | Every 12 weeks, up to 2 years
  Time from the first day of study treatment to the date of death due to any cause.
Best Overall Response | Every 12 weeks, up to 2 years
  The best response designation between the date of the first study treatment and the date of objectively documented progression or the date of subsequent anti-cancer therapy
Pharmacokinetic parameter: Cmax | Over the first 6 cycles (each cycle is 21 days) of patients treated with NP137 and enrolled during the Safety run in period
  Plasma peak concentration
Pharmacokinetic parameter: tmax | Over the first 6 cycles (each cycle is 21 days) of patients treated with NP137 and enrolled during the Safety run in period
  Time to reach the peak concentration
Pharmacokinetic parameter: AUCt | Over the first 6 cycles (each cycle is 21 days) of patients treated with NP137 and enrolled during the Safety run in period
  Area under the concentration-time curve from time zero to the last sample with the quantifiable concentration
Pharmacokinetic parameter: AUC∞ | Over the first 6 cycles (each cycle is 21 days) of patients treated with NP137 and enrolled during the Safety run in period
  Area under the concentration-time curve from time zero to infinity corresponding to the definite integral of a curve that describes the variation of a drug concentration in blood plasma as a function of time (drug exposure in plasma)
Pharmacokinetic parameter: CL | Over the first 6 cycles (each cycle is 21 days) of patients treated with NP137 and enrolled during the Safety run in period
  Clearance: volume of plasma from which NP137 is completely removed per unit time.
Pharmacokinetic parameter: t1/2 | Over the first 6 cycles of the patients Treated with NP137 and enrolled during the Safety run in period
  Terminal elimination half-life: time required for the amount of NP137 in the body to decrease by half.

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHRU BESANCON - Hopital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Primary Completion Date, Lille
  - Centre Léon Bérard, Lyon
  - Primary Completion Date, Marseille
  - ICM - Val d'Aurelle, Montpellier
  - Insitut de cancérologie de l'ouest, Nantes
  - Hopital de la Croix Saint Simon, Paris
  - Institut Curie (Site Saint Cloud), Paris
  - Institut Gustave Roussy, Paris
  - Aphp Cochin, Paris
  - Centre Eugène Marquis, Rennes
  - Institut claudius Regaud, Toulouse